CLINICAL TRIAL: NCT01158885
Title: Clofarabine With Cytarabine for MRD Positive Leukemia
Brief Title: Clofarabine With Cytarabine for Patients With Minimal Residual Disease Positive Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated for lack of accrual.
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2009-002
Record Dates: First submitted 2010-06-30; First posted 2010-07-08 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Minimal Residual Disease; Leukemia, Lymphoblastic, Acute; Leukemia, Myelogenous, Acute
Keywords: relapsed; relapse; refractory; Minimal Residual disease; MRD; MRD positive; MRD+; ALL; Acute lymphoblastic leukemia; AML; Acute myelogenous leukemia; Relapsed AML
MeSH Terms: conditions — Neoplasm, Residual; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Recurrence | interventions — Clofarabine; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): A maximum of two courses of the following regimen will be administered.
  * Clofarabine: 20 mg/m2/day intravenously (IV) over 2 hours (given at hours 0 to 2) on days 1 through 5.
  * Cytarabine intravenous: 1 gram/m2/day intravenously (IV) over 2 hours to be given 4 hours after the initiation of clofarabine on days 1 through 5.
  * Methotrexate: to be given intrathecally (IT) to all acute lymphoblastic leukemia (ALL) patients on day 1 at the dose defined by age.
  * Intrathecal (IT) cytarabine: is optional for acute myelogenous leukemia (AML) patients.
  Interventions: Drug: Clofarabine; Drug: Cytarabine intravenous; Drug: Methotrexate; Drug: Intrathecal (IT) Cytarabine

INTERVENTIONS:
Drug: Clofarabine — 20 mg/m2/day intravenously (IV) over 2 hours (given at hours 0 to 2) on days 1 through 5.
  Other Names: Clolar; CAFdA; Cl-F-ara-A
Drug: Cytarabine intravenous — 1 gram/m2/day intravenously (IV) over 2 hours to be given 4 hours after the initiation of clofarabine on days 1 through 5.
  Other Names: AraC; Cytosine arabinoside; Cytosar
Drug: Methotrexate — Methotrexate to be given intrathecally (IT) to all acute lymphoblastic leukemia (ALL) patients on day 1 at the dose defined by age below:
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  Other Names: MTX; Amethopterin
Drug: Intrathecal (IT) Cytarabine — Intrathecal (IT) cytarabine is optional for acute myelogenous leukemia (AML) patients.
  If intrathecal cytarabine is to be given, it must be given at least 72 hours but not more than 7 days prior to the initiation of intravenous cytarabine.
  Dose should be given according to age as defined below:
  * 30 mg for patients age 1-1.99
  * 50 mg for patients age 2-2.99
  * 70 mg for patients >3 years of age
  Other Names: AraC; Cytosine arabinoside; Cytosar

SUMMARY:
This study will test the ability of clofarabine + cytarabine to eliminate minimal residual disease (MRD) in acute myelogenous leukemia (AML) and acute lymphoblastic leukemia (ALL) patients whose bone marrows exhibit complete remission by morphology. The toxicity profile of this regimen will be evaluated in addition to toxicity experienced by patients who proceed to stem cell transplant. Overall length of remission will also be collected.

DETAILED DESCRIPTION:
Recent studies have demonstrated that even low levels of minimum residual disease (MRD) (>0.01% abnormal blasts) after aggressive re-induction therapy indicate a relatively poor outcome in relapsed acute lymphoblastic leukemia (ALL) patients, including those who proceed to allogeneic stem cell transplant (alloSCT). A similarly poor prognosis was seen in pediatric acute myelogenous leukemia patients with sub-morphologic disease prior to alloSCT. Studies to identify therapies that can eliminate persistent leukemia, have low toxicity profiles and can serve as a bridge to transplant are needed.

This study will test the ability of clofarabine + cytarabine to eliminate minimal residual disease (MRD) in acute myelogenous leukemia and acute lymphoblastic leukemia patients whose bone marrows exhibit complete remission by morphology. The toxicity profile of this regimen will be evaluated in addition to toxicity experienced by patients who proceed to stem cell transplant. Overall length of remission will also be collected.

ELIGIBILITY:
A. INCLUSION CRITERIA

1. Patients must be ≥1 and ≤ 21 years of age when enrolled onto this study.
2. Diagnosis

   * Patients must have a diagnosis of relapsed or refractory AML or ALL and,
   * Patient must have an M1 marrow based upon a recovered marrow with less than 5% blasts by conventional morphology and,
   * Patient must have minimal residual disease (MRD) detected by either multidimensional or conventional flow cytometry greater than 0.1% and less than 5% following any re-induction attempt and
   * Patients must be CNS 1.
3. Patient must have an ANC >500/μL off cytokine support for at least 24 hours and platelets >50,000 K/μL without platelet transfusion in the past seven days
4. Performance Level Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤16 years of age.
5. Patient must have adequate venous access.
6. Prior Therapy

   1. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
   2. At least 21 days must have elapsed from prior chemotherapy, at least 7 days must have elapsed since receiving biological therapy.
   3. It must be at least 45 days from any higher dose cytarabine therapy (>1 gm/ m2/day).
   4. Patients on steroid taper must be on less than 0.5mg/kg/day with plans to continue taper and discontinue the steroids.
7. Renal and Hepatic Function Patient must have adequate renal and hepatic functions as indicated by the following laboratory values:

   1. Patients must have a normal calculated creatinine clearance as calculated below:

      * Pediatric Population (age <18): Calculated creatinine clearance ≥ 90 ml/min/1.73m2 as calculated by the Schwartz formula for estimated glomerular filtration rate (GFR) where GFR (ml/min/1.73 m2) = k*Height (cm)/serum creatinine (mg/dl). k is a proportionality constant which varies with age and is a function of urinary creatinine excretion per unit of body size; 0.45 up to 12 months of age; 0.55 children and adolescent girls; and 0.70 adolescent boys.
      * Adult Population (age ≥18): Serum creatinine ≤1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black.
   2. Conjugated (direct) serum bilirubin ≤ 1.5 x ULN for age.
   3. Alanine transaminase (ALT) ≤ 2.5 × ULN for age.
   4. Alkaline phosphatase ≤ 2.5 × ULN for age.
   5. Serum amylase ≤ 1.5 ULN for age.
   6. Serum Lipase is ≤ ULN for age.
8. Patient must have a shortening fraction > 28% by echocardiogram or an ejection fraction > 50% by MUGA
9. Reproductive Function

   1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
   2. Female patients with infants must agree not to breastfeed their infants while on this study.
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.
10. Patient must agree to submission of blood and bone marrow for MPF assessment of MRD to TACL centralized lab.

B. EXCLUSION CRITERIA

Patients will be excluded if they meet any of the following criteria:

1. Patients with previous HSCT within previous 180 days.
2. Patients who have had prior treatment with clofarabine.
3. Patients with CNS2 or CNS 3 disease or bulky chloromatous disease.
4. Patients with Down Syndrome.
5. Patients with a previous history of veno-occlusive disease (VOD) or findings consistent with a diagnosis of VOD, defined as: conjugated serum bilirubin >1.4 mg/dL AND unexplained weight gain greater than 10% of baseline weight or ascites AND hepatomegaly or right upper quadrant pain without another explanation, OR reversal of portal vein flow on ultrasound, OR pathological confirmation of VOD on liver biopsy.
6. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
7. Use of investigational agents within 30 days of planned treatment on this protocol.
8. Patient is receiving or plans to receive concomitant chemotherapy, radiation therapy, immunotherapy or other anti-cancer therapy other than is specified in the protocol.
9. Pregnant or lactating patients.
10. Any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
11. Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy with the following exceptions:

    1. Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
    2. Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
12. Patient has active acute (greater than grade II) or active chronic extensive GVHD. Patients who are on a tapering dose of immunosuppressants will be permitted (tapering calcineurin inhibitor and/or less than 0.5 mg/kg/day of steroids).

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10-24 (Actual); Study Completion 2012-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blythe Thomson, MD, Study Chair — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Carolina-Levine Children's Hospital, Charlotte, North Carolina
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Clofarabine, Cytarabine, Methotrexate
  See detailed description in Interventions section.
Period: Treatment Course 1
Arm/Group | Single Arm
Started | 2
Completed | 2
Not Completed | 0
Period: Treatment Course 2
Arm/Group | Single Arm
Started (Neither of the patients that were treated on Treatment Course 1 were eligible to proceed to Course 2) | 0 (Neither of the patients that were treated on Treatment Course 1 were eligible to proceed to Course 2)
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Minimal Residual Disease (MRD)
Description: To be assessed in acute myelogenous leukemia (AML) and acute lymphoblastic leukemia (ALL) patients whose bone marrows exhibit complete remission by morphology. Patient's bone marrow will be evaluated for the amount of minimal residual disease (MRD) present after treatment on courses 1 and 2.
Time Frame: Sample collected between Days 22-36 of courses 1 and 2
Population: Study was closed prematurely and none of the patients treated were eligible for analysis of disease response.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients With Dose-Limiting Toxicity (DLT)
Description: Treatment related toxicities that preclude proceeding to HSCT by day 56 of the treatment course.
Time Frame: Beginning with the first dose of investigational product until day 56 of treatment course, an average of 1 year
Population: All patients treated on Treatment Course 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Occurrence of Toxicity During Hematopoietic Cell Transplant (HCT) for Patients Who Achieve Remission and Proceed to Transplant
Description: After the patient completes therapy on this protocol, data will continue to be collected regarding whether the patient proceeded to HCT. Toxicity and adverse event information will be collected.
Time Frame: Every 3 months for life following completion of protocol therapy.
Population: None of the patients treated on Treatment Course 1 proceeded to HCT. 1 patient upon completion of Treatment Course 1 proceeded with Bone Marrow Transplant and 1 patient was removed early from protocol treatment during Course 1 due to progressive disease.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 2 years
Description: The definition of AE and SAE used to collect adverse event information does not differ from the clinicaltrials.gov definitions.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Grade 4 Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=2)
Alanine aminotransferase (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Leukopenia NOS (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The study only enrolled two patients and closed early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days